CLINICAL TRIAL: NCT01730586
Title: Phase II Study of Abraxane in CIMP-High Colorectal Adenocarcinomas and Small Bowel Adenocarcinomas
Brief Title: Abraxane in CIMP-High Colorectal and Small Bowel Adenocarcinomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0776; NCI-2013-00077 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-10-26; First posted 2012-11-21 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Colorectal Cancer; Cancer of Gastrointestinal Tract
Keywords: Colorectal Cancer; Cancer of Gastrointestinal Tract; CIMP-high Colorectal Adenocarcinoma; Small Bowel Adenocarcinomas; Colorectal; Small bowel cancer; Abraxane; Nab-Paclitaxel; Paclitaxel (Protein-Bound); ABI-007
MeSH Terms: conditions — Colorectal Neoplasms; Gastrointestinal Neoplasms | interventions — Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abraxane (Experimental): Abraxane 220 mg/m2 administered by vein on Day 1. A cycle of therapy is defined as 21 days.
  Interventions: Drug: Abraxane

INTERVENTIONS:
Drug: Abraxane — 220 mg/m2 administered by vein on Day 1. A cycle of therapy is defined as 21 days.
  Other Names: Nab-Paclitaxel; Paclitaxel (Protein-Bound); ABI-007

SUMMARY:
The goal of this clinical research study is to learn if abraxane can help to control colorectal and/or small bowel cancer. The safety of this drug will also be studied.

Abraxane is designed to block cancer cells from dividing, which may cause them to die.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive the study drug in 21-day study cycles.

You will receive abraxane by vein over about 30 minutes on Day 1 of each cycle.

Study Visits:

On Day 1 of all cycles, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and blood pressure.
* You will be asked about any drugs you may be taking and about any symptoms or side effects you may be having.
* Your performance status will be recorded.
* Blood (about 2 tablespoons) will be drawn for routine tests.

At the end of every 3rd cycle (Cycles 3, 6, 9) and so on:

°You will have a CT or MRI scan of your chest, abdomen, and pelvis to check the status of the disease. If at any point the scans show the disease appearing to get better, you will have another scan 2 cycles later.

Length of Treatment:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if you have intolerable side effects, if the study is stopped, or if you are unable to follow study instructions.

Your participation on the study will be over after the follow-up period.

End-of-Treatment Visit:

Within 10 days after you stop taking the study drug, you will have an end-of-treatment visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and blood pressure.
* You will be asked about any drugs you may be taking and about any symptoms or side effects you may be having.
* Your performance status will be recorded.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* If one has not been performed in the previous 4 weeks, you will have a CT or MRI scan of your chest, abdomen, and pelvis to check the status of the disease.

Follow-Up:

The study staff will ask about any symptoms or side effects you may be having during the 30 days after your last dose of the study drugs. The study staff may ask you by phone or at the time of a routine clinic visit. If the study staff contacts you by phone, the phone call should last about 15-30 minutes.

If you leave the study for any reason other than the disease getting worse, you will have a CT or MRI scan of your chest, abdomen, and pelvis to check the status of the disease every 12 weeks unless you start receiving other treatment.

The study staff will also review your medical records and/or contact you to check the status of the disease every 3 months after you stop receiving the study drug. If you are contacted by phone, each phone call should take about 5 minutes.

This is an investigational study. Abraxane is FDA approved and commercially available for the treatment of breast cancer. It is not FDA approved for the treatment of colorectal or small bowel cancer. The use of abraxane in patients with colorectal cancer or small bowel cancer is investigational.

Up to 35 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histologically or cytologically confirmed colorectal adenocarcinoma or small bowel adenocarcinoma
2. Metastatic disease documented on diagnostic imaging studies with measurable disease per RECIST version 1.1.
3. Refractory disease defined as: a) prior treatment with fluoropyrimidine, oxaliplatin, irinotecan, and anti-epidermal growth factor receptor (EGFR) therapy if Kirsten rat sarcoma (KRAS) wildtype for colorectal adenocarcinoma and; b) prior treatment with fluoropyrimidine and oxaliplatin for small bowel adenocarcinoma.
4. Colorectal adenocarcinoma patients must be known to have CpG island methylator phenotype. CIMP-high phenotype will be defined as hypermethylation at 2 or more of the 6 methylation-specific PCR markers (hMLH1, P16, P14, MINT1, MINT2, and MINT31).
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
6. Adequate organ function including: a) Absolute neutrophil count (ANC) =/>1,500cells/mm^3; b) Platelets =/>100,000/ul; c) Hemoglobin >9.0 g/dL; d) Total bilirubin =/<1.5mg/dL In patients with known Gilbert's syndrome, direct bilirubin =/<1.5 x upper limit of normal (ULN) will be used as organ function criteria, instead of total bilirubin; e) AST and ALT < 2.5 x ULN; f) Alkaline phosphatase <2.5x ULN; g) Creatinine <1.5 gm/dL.
7. Negative serum or urine pregnancy test in women with childbearing potential (WOCBP) defined as not post-menopausal for 12 months or no previous surgical sterilization, within one week prior to initiation of treatment. WOCBP must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of study drug to minimize the risk of pregnancy.
8. A male subject of fathering potential must use an adequate method of contraception to avoid conception throughout the study and for up to 12 weeks after the last dose of study drug to minimize the risk of pregnancy. If the partner is pregnant or breastfeeding, the subject must use a condom.
9. Patients must sign an Informed Consent and Authorization indicating that they are aware of the investigational nature of this study and the known risks involved.
10. Patient is =/>18 years of age on the day of consenting to the study.

Exclusion Criteria:

1. Peripheral neuropathy of grade 2 or greater by Common Terminology Criteria for Adverse Events (CTCAE) 4.0. In CTCAE version 4.0 grade 2 sensory neuropathy is defined as "moderate symptoms; limiting instrumental activities of daily living (ADLs)".
2. Prior treatment with taxane therapy for either colorectal cancer or small bowel adenocarcinoma.
3. Chemotherapy or any other investigational agents within 14 days of first receipt of study treatment, or major surgery within 28 days of first receipt of study treatment, or palliative radiation within 7 days of first receipt of study treatment.
4. Concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study such as unstable angina, myocardial infarction within 6 months, unstable symptomatic arrhythmia, uncontrolled diabetes, serious active or uncontrolled infection.
5. Pregnancy (positive pregnancy test) or lactation.
6. Patients with carcinomatous meningitis.
7. Known central nervous system (CNS) disease, except for treated brain metastasis. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Overman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: November 2012 to October 2015. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Abraxane: Abraxane 220 mg/m^2 intravenously on Day 1 of 21 day cycle.
Period: Overall Study
Arm/Group | Abraxane
Started | 34
Completed | 21
Not Completed | 13
Not completed — Progressive Disease | 2
Not completed — Inadequate Trial | 8
Not completed — Adverse Event | 2
Not completed — Hospice | 1

BASELINE CHARACTERISTICS:
Arm/Group | Abraxane
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 59 [34 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 34
Colorectal Cancer Diagnosis [Count of Participants; unit: Participants] — Histologically or cytologically confirmed colorectal adenocarcinoma (CpG island methylator phenotype (CIMP-high)) or small bowel adenocarcinoma
  Participants
    Small Bowel Adenocarcinoma (SBA) | 13
    CIMP-high Colorectal Cancer (CRC) | 21

OUTCOME MEASURES:

1. Primary Outcome: Response Rate in CIMP-High Colorectal Cancer and Small Bowel Adenocarcinoma (SBA)
Description: Evaluated using Response Evaluation Criteria In Solid Tumors (RECIST) criteria (version 1.1, 2009): Complete Response (CR): Disappearance all lesions including normalization of elevated tumor marker level; Pathological lymph nodes reduction in short axis to <10 mm. Partial Response (PR): >30% decrease sum longest diameters (LD) of lesions reference baseline sum LD. Progressive Disease (PD): >20% increase (absolute increase >5 mm) in sum LD measured lesions references smallest sum LD, and appearance new lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference smallest sum LD. After a tumor demonstrates a tumor response (partial or complete), confirmation of the response obtained by a second evaluation to be performed 2 cycles later (+/- 1week) [second tumor assessment not <4 weeks from response observed]. Assessed via computed tomography (CT) of the chest, abdomen, and pelvis.
Time Frame: Assessed at 21 day cycle; Restaging done every 3 cycles
Population: In the CIMP-CRC arm 15 participants were considered efficacy evaluable [Of 21 treated, 6 participants were withdrawn due to toxicity (2) and due to clinical progression (4)], and three were not evaluable in SBA arm.
Measure: Count of Participants; unit: Participants
Groups:
- CIMP-high Colorectal Cancer; Small Bowel Adenocarcinoma (SBA): Abraxane 220 mg/m^2 intravenously on Day 1 of 21 day cycle.
Arm/Group | CIMP-high Colorectal Cancer | Small Bowel Adenocarcinoma (SBA)
Number analyzed (Participants) | 15 | 10
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 2
  Stable Disease | 3 | 3
  Progressive Disease | 12 | 5

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: The length of time during and after the treatment a participant lives without disease progression. Time to progression functions estimated using the Kaplan-Meier method. Participants who drop out of the study included in the time to event data analysis as "censored data".
Time Frame: Assessed at first cycle (21 days), up to 12 months
Population: For progression-free survival, the intent-to-treat analysis performed using all available participants.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Small Bowel Adenocarcinoma: Abraxane 220 mg/m^2 intravenously on Day 1 of 21 day cycle.
Arm/Group | CIMP-high Colorectal Cancer | Small Bowel Adenocarcinoma
Number analyzed (Participants) | 21 | 13
Months | 2.1 [1.7 to 2.5] | 3.2 [2.6 to 3.8]

ADVERSE EVENTS:
Time Frame: Through Day 30 (Day 28 to Day 45 allowed) following the last dose of study drug or until resolution or stabilization of the toxicity or start of another treatment regimen, up to 3 years
Arm/Group | Abraxane
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 20/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abraxane (N=34)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 6
Jejunal obstruction (Gastrointestinal disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Infection, Other - perirectal abcess (Infections and infestations) | 1
Rectal pain (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Hypotension (Vascular disorders) | 2
Confusion (Psychiatric disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abraxane (N=34)
Abdominal distension (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 9 (18)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (4)
Alkaline phosphatase increased (Investigations) | 7 (7)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 26 (26)
Anemia (Blood and lymphatic system disorders) | 12 (15)
Anorexia (Metabolism and nutrition disorders) | 9 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (20)
Ascites (Gastrointestinal disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Blood bilirubin increased (Investigations) | 3 (5)
Blurred vision (Eye disorders) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Concentration impairment (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 5 (6)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (19)
Dizziness (Nervous system disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Edema face (General disorders) | 2 (2)
Edema limbs (General disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Eye disorders (Eye disorders) | 1 (1)
Fatigue (General disorders) | 21 (39)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Fever (General disorders) | 5 (5)
Flatulence (Gastrointestinal disorders) | 2 (2)
Flu like symptoms (General disorders) | 2 (2)
Flushing (Vascular disorders) | 4 (9)
Gait disturbance (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - (Other) (Gastrointestinal disorders) | 1 (3)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (5)
Hematoma (Vascular disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (7)
Hypotension (Vascular disorders) | 3 (4)
Hypothyroidism (Endocrine disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2)
Infections and infestations - (Other) (Infections and infestations) | 2 (4)
Insomnia (Psychiatric disorders) | 3 (5)
Investigations - (Other) (Investigations) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 3 (3)
Malaise (General disorders) | 3 (4)
Menorrhagia (Reproductive system and breast disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 7 (8)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (28)
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 14 (24)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (6)
Pain (Musculoskeletal and connective tissue disorders) | 7 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (9)
Platelet count decreased (Investigations) | 5 (8)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (6)
Rectal pain (Gastrointestinal disorders) | 1 (4)
Reproductive system and breast disorders - (Other) (Reproductive system and breast disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin and subcutaneous tissue disorders - (Other) (Skin and subcutaneous tissue disorders) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Soft tissue infection (Infections and infestations) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (12)
Weight loss (Investigations) | 5 (5)
White blood cell decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes